CLINICAL TRIAL: NCT02817594
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in The Netherlands (3DUTCH)
Brief Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program in Patients With Chronic Hepatitis C
Acronym: 3DUTCH
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-788
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Paritaprevir/r - Ombitasvir, ± Dasabuvir; Sustained Virological Response; Observational Study; Chronic Hepatitis C genotype 1; Chronic Hepatitis C genotype 4
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
  The prescription of treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
The interferon-free combination regimen of paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) for the treatment of chronic hepatitis C (CHC) has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well controlled conditions.

This observational study is the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in the Netherlands in a clinical practice patient population.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female participants with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with the current local label.
* If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy).
* Participants must voluntarily sign and date informed consent prior to inclusion into the study

Exclusion Criteria:

* Patients participating or intending to participate in a concurrent interventional therapeutic trial.
* Unable to complete the questionnaires due to cognitive impairment or lack of any kind of cognitive competence, as to be judged by the healthcare professional who is treating the patient.
* Unable to complete the questionnaires due to language incompetence.
* Unable to voluntarily sign and date the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients chronically infected with HCV, receiving the interferon-free ABBVIE REGIMEN will be offered the opportunity to participate in this study during a routine clinical visit at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (9):
- Netherlands (9):
  - Albert Schweitzer Ziekenhuis /ID# 152597, Dordrecht, South Holland
  - Noordwest Ziekenhuisgroep /ID# 152604, Alkmaar
  - Duplicate_Onze Lieve Vrouwe Gasthuis /ID# 152600, Amsterdam
  - Universitair Medisch Centrum Groningen /ID# 152596, Groningen
  - Leids Universitair Medisch Centrum /ID# 154637, Leiden
  - Radbound University Medical Ce /ID# 152598, Nijmegen
  - Erasmus Medisch Centrum /ID# 154635, Rotterdam
  - Maasstad Ziekenhuis /ID# 152592, Rotterdam
  - Universitair Medisch Centrum Utrecht /ID# 152595, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants chronically infected with hepatitis C virus (HCV) were enrolled at 9 centers in the Netherlands.
Pre-assignment Details: Participants were prescribed the interferon-free combination regimen of paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) at the discretion of the physician in accordance with local clinical practice and label.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Started | 51
Received Treatment | 50
Completed (Completed defined as having an HCV RNA assessment performed at least 10 weeks post-treatment) | 48
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Not completed — Did Not Receive Treatment | 1

BASELINE CHARACTERISTICS:
Population: Treated participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks, according to HCV genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hepatitis C Virus Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 9
  Genotype 1b | 34
  Genotype 4a | 2
  Genotype 4d | 1
  Genotype 4n | 1
  Genotype 4r | 1
  Genotype 4, Subtype Unknown | 2
Cirrhosis status [Count of Participants; unit: Participants]
  No cirrhosis | 40
  Transition to cirrhosis | 4
  Cirrhosis | 6
Years Since Diagnosis of HCV Infection [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 49
    (all) | 12.3 (12.41)
HCV Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log10 IU/mL] — Population: Enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) with non-missing RNA data.
  log10 IU/mL
    number analyzed (Participants) | 47
    (all) | 5.98 (0.925)
Assigned Treatment Regimen [Count of Participants; unit: Participants] — Treatment regimen was assigned by the physician according to local practice and label. Participants could receive two (paritaprevir/ritonavir and ombitasvir) or three (paritaprevir/ritonavir, ombitasvir, and dasabuvir) direct-acting antiviral (DAA) drugs with or without ribavirin for 12 or 24 weeks.
  Participants
    2 DAA without RBV for 12 weeks | 2
    2 DAA with RBV for 12 weeks | 4
    3 DAA without RBV for 12 weeks | 34
    3 DAA with RBV for 12 weeks | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug. Participants with missing HCV RNA were counted as virological failure.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The Core Population, defined as enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks according to HCV genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 48
percentage of participants | 89.6 [77.8 to 95.5]

2. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen)
Population: The Core Population defined as enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 48
percentage of participants | 95.8 [86.0 to 98.8]

3. Secondary Outcome: Percentage of Participants With Sufficient Follow-up Who Achieved Sustained Virological Response 12 Weeks Post-treatment
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
  The Core Population with sufficient follow-up data regarding SVR12 included all core population participants who
  * had evaluable HCV RNA data ≥ 70 days after the last actual dose of the ABBVIE REGIMEN
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 70 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The Core Population with sufficient follow-up data regarding SVR12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 47
percentage of participants | 91.5 [80.1 to 96.6]

4. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen) and up to 24 weeks after the end of treatment.
Population: The Core Population with VR at EOT and who completed treatment, and had ≥ 1 HCV RNA measurement ≥ 70 days post-treatment or were a treatment failure between EOT and day 70.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 44
percentage of participants | 6.8 [2.3 to 18.2]

5. Secondary Outcome: Percentage of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 12 or 24 weeks (depending on the treatment regimen)
Population: The Core Population with virological response on-treatment and with at least one on-treatment measurement thereafter (including EOT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 8
percentage of participants | 0.0 [0.0 to 32.4]

6. Secondary Outcome: Percentage of Participants in Each Non-response Category 12 Weeks Post-treatment
Description: SVR12 non-response was categorized according to the following:
  * On-treatment virologic failure (breakthrough [at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥ 50 IU/mL]);
  * Relapse, defined as HCV RNA < 50 IU/mL at EOT followed by HCV RNA ≥ 50 IU/mL post-treatment in patients who completed treatment (not more than 7 days shortened);
  * Premature treatment discontinuation with no on-treatment virologic failure;
  * Missing SVR12 data and/or none of the above criteria.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The Core Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 48
Participants
  On-treatment virologic failure | 0
  Relapse | 3
  Premature treatment discontinuation | 1
  None of the above criteria | 1

7. Secondary Outcome: Percentage of the Direct Acting Antiviral (DAA) Dose Taken in Relation to the Target Dose of DAA
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: The Core Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 48
Participants
  > 105 % | 1
  > 95% to ≤ 105% | 41
  > 80% to ≤ 95% | 2
  > 50% to ≤ 80% | 2
  ≤ 50% | 1
  Missing | 1

8. Secondary Outcome: Percentage of the Ribavirin Dose Taken in Relation to the Target Dose of Ribavirin
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: The Core Population who were prescribed ribavirin.
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 14
Participants
  > 105% | 1
  > 95% to ≤ 105% | 11
  > 80% to ≤ 95% | 0
  > 50% to ≤ 80% | 0
  ≤ 50% | 2

9. Secondary Outcome: Percentage of Ribavirin (RBV) Treatment Days in Relation to the Target Number of Ribavirin Treatment Days
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: The Core Population who were prescribed ribavirin.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 14
percentage of days | 96.0 (19.62)

10. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, or Pregnancies
Time Frame: From first dose of study drug through 30 days after last dose (16 weeks).
Population: The Safety Population, defined as all enrolled participants who received at least one dose of the ABBVIE regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 50
Participants
  Any adverse event | 32
  Serious adverse event | 2
  Pregnancy | 0

11. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score by applying country-specific weights.The range for EQ-5D-5L index score is 0 to 1 where '0' is defined as a health state equivalent to being dead and '1' is full health.The higher the score the better the health status.
Time Frame: Baseline, end of treatment (week 12 or 24 depending on the treatment regimen), and at 12 and 24 weeks after end of treatment
Population: The Core Population with available data at baseline and each time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 43
units on a scale
  End of treatment: number analyzed (Participants) | 40
  End of treatment | 0.000 [-0.131 to 0.015]
  12 weeks after end of treatment: number analyzed (Participants) | 36
  12 weeks after end of treatment | 0.000 [-0.082 to 0.096]
  24 weeks after end of treatment: number analyzed (Participants) | 24
  24 weeks after end of treatment | 0.000 [-0.084 to 0.115]

12. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status with a separate visual analog scale (VAS).
  The VAS assesses overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: as for outcome 11
Population: The Core Population with available data at baseline and each time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 44
units on a scale
  End of treatment: number analyzed (Participants) | 42
  End of treatment | 0.0 [-15.0 to 5.0]
  12 weeks after end of treatment: number analyzed (Participants) | 38
  12 weeks after end of treatment | 0.0 [-10.0 to 11.0]
  24 weeks after end of treatment: number analyzed (Participants) | 25
  24 weeks after end of treatment | 0.0 [-10.0 to 10.0]

13. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Absenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Absenteeism indicates the percentage of work time missed due to health problems.
Time Frame: as for outcome 11
Population: The Core Population who were employed and with available data at baseline and each time point.
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 17
percent impairment
  End of treatment: number analyzed (Participants) | 14
  End of treatment | 0.0 [0.0 to 0.0]
  12 weeks after end of treatment: number analyzed (Participants) | 12
  12 weeks after end of treatment | 0.0 [0.0 to 0.0]
  24 weeks after end of treatment: number analyzed (Participants) | 10
  24 weeks after end of treatment | 0.0 [0.0 to 42.9]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after last dose (16 weeks).
Groups:
- 2 DAA: Participants received paritaprevir/ritonavir and ombitasvir for 12 weeks.
- 2 DAA + RBV: Participants received paritaprevir/ritonavir and ombitasvir plus ribavirin for 12 weeks.
- 3 DAA: Participants received paritaprevir/ritonavir, ombitasvir, dasabuvir, without ribavirin, for 12 weeks.
- 3 DAA + RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir plus ribavirin for 12 weeks.
Arm/Group | 2 DAA | 2 DAA + RBV | 3 DAA | 3 DAA + RBV
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 1/34 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 2/34 | 0/10
Other Adverse Events (participants affected / at risk) | 1/2 | 1/4 | 22/34 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA (N=2) | 2 DAA + RBV (N=4) | 3 DAA (N=34) | 3 DAA + RBV (N=10)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA (N=2) | 2 DAA + RBV (N=4) | 3 DAA (N=34) | 3 DAA + RBV (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 12 (12) | 7 (7)
SENSE OF OPPRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6) | 3 (3)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02817594/SAP_000.pdf
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT02817594/Prot_001.pdf